CLINICAL TRIAL: NCT06051097
Title: Relationship Between Metabolic Syndrome and Obstructive Sleep Apnea
Brief Title: Metabolic Syndrome and Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Kamal Ibrahim Hassan, Assistant Professor of pulmonology, Cairo University
Other Study IDs: MS-258-2022
Record Dates: First submitted 2023-09-04; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Sleep Apnea; Metabolic Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes; Metabolic Syndrome | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sampling for lipid profile and HBAIC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA with metabolic syndrome: sleep study
  Interventions: Diagnostic Test: sleep study
- OSA without metabolic syndrome: sleep study
  Interventions: Diagnostic Test: sleep study

INTERVENTIONS:
Diagnostic Test: sleep study — over-night polysomnography

SUMMARY:
Background:Metabolic syndrome is a disorder characterized by abdominal obesity,hypertension,increased triglycerides ,decreased HDL cholesterol and increased blood glucose. Accumulating evidence strongly indicates that insulin resistance and an increased amount of abdominal fat are the pathogenic factors for the characteristics of metabolic syndrome. Studies indicate that sleep apnea may be a manifestation of the metabolic syndrome.

Subjects and methods:This study was conducted in the pulmonology department at kasrelainy hospital. It included 80 patients who came to the sleep lab unit for polysomnography. Each patient was subjected to full history taking including(sex,age,smoking history,presence of diabetes or hypertension),thorough clinical examination with emphasis on waist, neck&hip circumference and blood pressure measurements,Laboratory investigations including :Lipid profile& Diabetic profile(HBA1C).In addition to ESS and stop bang score questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilled the criteria of OSA ( obstructive sleep apnea) in the form of symptoms suggestive of OSA (daytime sleepiness/daytime fatigue/headache/snoring)and with AHI ( apnea-hyponea index) ≥5.

Exclusion Criteria:

1. Cerebro-vascular accident within the preceding 30 days.
2. Patients on sedatives.
3. Patients on anti-psychotics

Ages: 22 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted in the pulmonology department at kasrelainy hospital.Itincluded 80 patients who came to the sleep lab unit for polysomnography.Each patient was subjected to full history taking including(sex,age,smoking history,presence of diabetes or hypertension),thorough clinical examination with emphasis on waist, neck & hip circumference and blood pressure measurements,Laboratory investigations including: Lipid profile&Diabetic profile(HBA1C).In addition to ESS and stop-bang score questionnaire
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Predictors of metabolic syndrome among OSA patients | 6 months
  evaluation of factors related to occurrence of metabolic syndrome in OSA such as age(in years),weight in kilograms(kg) and height in meters (m) will not be measured separately but combined to assess BMI( weight in kg/ height in m2) and oxygen saturation (O2%), evaluation of polysomnographic data and laboratory tests in the form of lipid profile in (mg/dl) and HBA1C (g/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy school of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No